CLINICAL TRIAL: NCT04147520
Title: Reducing Hazardous Alcohol Use in Social Networks Using Targeted Intervention: 21 Rising
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1810002247; 2R01AA023522 (NIH)
Record Dates: First submitted 2019-10-23; First posted 2019-11-01 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Alcohol Drinking; Alcohol; Harmful Use
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Motivational Interview (Active Comparator): Single-session in person conversation focusing on risks associated with alcohol use.
  Interventions: Behavioral: Brief Motivational Interview
- Natural History Control (No Intervention): No contact.

INTERVENTIONS:
Behavioral: Brief Motivational Interview — Single (60 min) session discussion of alcohol use and associated experiences.
  Arms: Brief Motivational Interview

SUMMARY:
The primary goal of this study is to determine whether change in alcohol use among college students can be transmitted through social network ties to other members in the network. Members of one college class at a northeastern university will be enrolled in a longitudinal study in which they will provide self-reported behavioral information and information about their social ties to others in their college class. A subset of heavy drinking participants will be asked to meet in person to complete an interview about their alcohol use - called a Brief Motivational Interview. There is evidence that this sort of interview can reduce harmful alcohol use. The investigators expect that following the Brief Motivational Interview others in their friendship clusters will show reduced harm associated with alcohol use as well.

ELIGIBILITY:
Inclusion Criteria:

• Must be a member of the class of 2021 or 2021.5 at the site university

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1475 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol use | At each follow up, measure average drinks per week in the past 30 days
  Average number of drinks per week in the past 30 days
Average number of alcohol consequences in the past 30 days | At each follow up, measure count of alcohol consequences in the past 30 days
  Count of alcohol consequences in the past 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Barnett, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
There is concern that with information in the dataset, including social ties, individuals could be re-identified.